CLINICAL TRIAL: NCT06387381
Title: 68Ga-PSFA PET Imaging in Patients With PSMA/FAP Positive Disease
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: First Affiliated Hospital of Chongqing Medical University (Other)
Responsible Party: Principal Investigator, Xiaoyang Zhang, Principal Investigator, First Affiliated Hospital of Chongqing Medical University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CYYY-KY-2024-048-01
Record Dates: First submitted 2024-04-24; First posted 2024-04-29 (Actual); Last update posted 2025-06-04 (Actual); Status verified 2025-05

CONDITIONS: PSMA; FAP; Positron-Emission Tomography

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- 68Ga-PSFA (Experimental): Patients will receive a single administration of 68Ga-PSFA.
  Interventions: Drug: 68Ga-PSFA

INTERVENTIONS:
Drug: 68Ga-PSFA — Each subject receives a single intravenous injection of 68Ga-PSFA.

SUMMARY:
As a new dual receptor (PSMA and FAP) targeting PET radiotracer, 68Ga-PSFA is promising as an excellent imaging agent applicable to PSMA/FAP positive diseases. In this research, we investigate the safety, biodistribution and potential usefulness of 68Ga-PSFA positron emission tomography (PET) for the diagnosis of lesions in PSMA/FAP positive diseases.

ELIGIBILITY:
Inclusion Criteria:

1. At least 18 years of age.
2. Signed informed consent.
3. Patients with suspected or newly diagnosed or previously malignant disease, with either PSMA or FAP positive expression (supporting evidence may include MRI, CT, and pathology report, etc).

Exclusion Criteria:

1. Patients with non-malignant disease.
2. Patients with pregnancy.
3. The inability or unwillingness of the research participant, parent or legal representative to provide written informed consent.
4. Known or expected hypersensitivity to 68Ga-PSFA or any of its components.
5. Any serious medical condition or extenuating circumstance which the investigator feels may interfere with the procedures or evaluations of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-05-20 (Actual); Primary Completion 2025-04-30 (Actual); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Diagnostic efficacy | 15 days
  The sensitivity, specificity, and accuracy of 68Ga-PSFA PET

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Chongqing Medical University, Chongqing, Chongqing Municipality, China

REFERENCES:
- [Derived] Wang X, Zhang X, Zhang X, Guan L, Gao X, Xu L, Pang H, Du J, Zhang J, Cui M. Design, preclinical evaluation, and first-in-human PET study of [68Ga]Ga-PSFA-01: a PSMA/FAP heterobivalent tracer. Eur J Nucl Med Mol Imaging. 2025 Feb;52(3):1166-1176. doi: 10.1007/s00259-024-06965-7. Epub 2024 Nov 9. PMID 39520516